CLINICAL TRIAL: NCT05130931
Title: Impact of a Conservative Treatment in the Waiting List for Carpal Tunnel Syndrome Surgery: Pilot Study.
Brief Title: Impact of a Conservative Treatment in the Waiting List for Carpal Tunnel Syndrome Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Mar Hernández Secorún, Teaching Assistant and PhD student, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHS1
Record Dates: First submitted 2021-10-29; First posted 2021-11-23 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal Conservative Treatment (Experimental)
  Interventions: Other: Multimodal conservative treatment
- Standard healthcare. (No Intervention)

INTERVENTIONS:
Other: Multimodal conservative treatment — 15 min of Pain education + 20 min of Specific mobilization of the forearm musculature, pronator teres, tendons of the palmar flexors of the wrist and fingers, transverse carpal ligament and palmar fascia through manual mobilization assisted by Diacutaneous Fibrolysis technique + 10min of self-management and explanation of home-based exercise.
  3 sessions of 45 minutes will be taken to perform this protocol and the patient will be shown a self-treatment to be performed 3-5 times a day. The protocol will be carried out over 3 weeks (1 session per week).
  Arms: Multimodal Conservative Treatment

SUMMARY:
STC is considered one of the most prevalent peripheral neuropathy of the upper quadrant. Systematic review shows that conservative treatment is effective for treatment of CTS. In Spain, most patients diagnosed by CTS are included in surgery list without considering conservative treatment as first option or providing drugs or night splint . However, surgical treatment is not always necessary for these patients, and waiting list delays can lead to aggravation of patients' symptoms.

Researches believe that performing a conservative treatment including diacutaneous fibrolysis on carpal tunnel syndrome patients, could reduce waiting surgery list, reduce the cost-effectiveness rate of the surgical process and improve patient's satisfaction and clinical findings. In addition, patients of any level of severity and with systemic pathology will be included to define which patients would benefit from surgical treatment and which from physiotherapeutic treatment.

The aim is to find out the impact of a multimodal physiotherapy treatment in patients with Carpal Tunnel Syndrome (CTS) on the patient and the Aragonese Health System.

A randomized controlled clinical trial will be performed. First a pilot study will be carried out. Patients with carpal tunnel syndrome included on waiting surgery list of Miguel Servet Hospital will be recruited. They will be randomized into a control group (staying in waiting list and performing healthcare standard) and into an experimental group (3 sessions of 45 min of diacutaneous fibrolysis and homebased treatment). Different outcomes will be assessed at pre-treatment, at the end of treatment, 3 and 6 months later.

ELIGIBILITY:
Inclusion:

* Have been diagnosed with Carpal Tunnel Syndrome (CTS) after the electrophysiological test at the neurophysiology service of the Miguel Servet Hospital in Zaragoza and be on the waiting list for CTS surgery.
* Have experienced symptoms for more than two months.
* Have sufficient comprehension and communication skills to communicate their symptoms and to fill in the questionnaires.
* Ability to maintain supine and lateral decubitus without causing symptoms or altering the patient's condition.
* Accept and give consent to participate voluntarily in the study.

Exclusion:

* Previous carpal tunnel surgery on the same limb.
* History of trauma on the upper limb which CTS may be associated, other musculoskeletal or neurological pathologies affecting the upper limb (e.g., cervical radiculopathy).
* Pregnancy, due to the influence of fluid retention in the cause of CTS, remitting spontaneously after childbirth, breastfeeding or up to 3 years after these episodes.
* Present physical contraindications (red flags) in general that contraindicate physical treatment such as: trauma, malignancy, inflammation, infection, fever... or psychological contraindications (yellow flags) that may have a marked effect on the results of treatment.
* Present specific physical contraindications that contraindicate diacutaneous fibrolysis treatment, such as ulcerations and skin alterations.
* Have specific contraindications that contraindicate surgical intervention such as taking anticoagulants or antiplatelet agents.
* Having received a steroid injection in the previous 6 months or interventions on the CTS in the previous 3 months.
* Pending trial or litigation related to CTS.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Change in nocturnal symptoms intensity (VAS) | Change between baseline, post-treatment, 3 months after, 6 months after
  The Visual Analog Scale is a unidimensional measure of symptoms intensity. Is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (nocturnal symptoms) orientated from the left (worst) to the right (best). Nocturnal sumptoms were measured in the last 3 days.
Change in pain intensity (VAS) | Change between baseline, immediate before and after each session, post-treatment, 3 months after, 6 months after
  The Visual Analog Scale is a unidimensional measure of symptoms intensity. Is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (pain) orientated from the left (worst) to the right (best). Pain was measured in the last 3 days and currently.
Change in paresthesia intensity (VAS) | Change between baseline, immediate before and after each session, post-treatment, 3 months after, 6 months after
  The Visual Analog Scale is a unidimensional measure of symptoms intensity. Is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (paresthesia) orientated from the left (worst) to the right (best). Paresthesia was measured in the last 3 days and currently.
Change in BCTQ | Change between baseline, post-treatment, 3 months after, 6 months after
  The Boston Carpal Tunnel Questionnaire (BCTQ) is a disease-specific measure of self-reported symptom severity and functional status. It is frequently used in the reporting of outcomes from trials into interventions for carpal tunnel syndrome.
Change in DASH questionnaire | Change between baseline, post-treatment, 3 months after, 6 months after
  The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.

SECONDARY OUTCOMES:
Change in NRS | The Numeric Rating Scale is a one-dimensional measure of symptoms intensity in adults. In our study, it was used to quantify the intensity of other symptoms present. It is a segmented numeric version of the visual analog scale (VAS) in which a respondent
  Change between baseline, post-treatment, 3 months after, 6 months after
Change in Katz's Diagram | Change between baseline, post-treatment, 3 months after, 6 months after
  Katz hand diagram is a drawing made by a patient of symptoms such as numbness, tingling, or pain affecting the hand and fingers. The drawing is a useful means of eliciting symptoms that suggest carpal tunnel syndrome.
Change in MOS Sleep Scale | Change between baseline, post-treatment, 3 months after, 6 months after
  The Medical Outcomes Study Sleep Scale (MOS-Sleep) includes 12 items assessing sleep disturbance, sleep adequacy, somnolence, quantity of sleep, snoring, and awakening short of breath or with a headache.
Change in SF-36 | Change between baseline, post-treatment, 3 months after, 6 months after
  The 36-Item Short Form Survey (SF-36) is an oft-used, well-researched, self-reported measure of health.
Change in TSK | Change between baseline, post-treatment, 3 months after, 6 months after
  The Tampa Scale of Kinesiophobia (TSK) is a 17 item scale originally developed to measure the fear of movement related to chronic lower back pain.
Change in ULTT | Change between baseline, immediate before and after each session, post-treatment, 3 months after, 6 months after
  The Upper Limb Tension Test is performed to assess mechanosensitivity of median nerve. Range of movement, symptom's location, symptoms response and structural differentiation were assessed.
Change in Strength | Change between baseline, post-treatment, 3 months after, 6 months after
  Pinch and grip strength were assessed by a manual dynamometer to evaluate forearm, hand and fingers muscle strength.
Change in SWMT | Change between baseline, immediate before and after each session, post-treatment, 3 months after, 6 months after
  The Semmes-Weinstein monofilament test (SWMT) is a clinical widely used test to quantify the sensibility in patients with Carpal Tunnel Syndrome (CTS).
Change in Neuropen | Change between baseline, post-treatment, 3 months after, 6 months after
  The Neuropen combines an interchangeable 10 g monofilament for cutaneous pressure assessment, and a calibrated sterile Neurotip for assessing pain sensation.
Change in PGI-I | Change between post-treatment, 3 months after, 6 months after
  The Patient Global Impression of Improvement (PGI-I) is a global index that may be used to rate the response of a condition to a therapy (transition scale).

OTHER OUTCOMES:
NCV | Baseline
  Neural conduction velocity (NCV) test is used to assess nerve damage and dysfunction. It allows classification of the severity of the patient's dysfunction on mild, moderate or severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health of Science, University of Zaragoza, Zaragoza, Aragon, Spain